CLINICAL TRIAL: NCT02425722
Title: Phase II Study of ASP0456 - A Double-blind, Placebo-controlled, Parallel-group, Comparative Study in Patients With Chronic Constipation (Not Including Constipation Due to Organic Diseases)
Brief Title: A Study to Evaluate Dose Responses of Efficacy and Safety of ASP0456 in Patient With Chronic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0456-CL-1021
Record Dates: First submitted 2015-04-07; First posted 2015-04-24 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Chronic Constipation
Keywords: linaclotide; ASP0456; chronic constipation
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- ASP0456 0.0625mg (Experimental): oral
  Interventions: Drug: ASP0456
- ASP0456 0.125mg (Experimental): oral
  Interventions: Drug: ASP0456
- ASP0456 0.25mg (Experimental): oral
  Interventions: Drug: ASP0456
- ASP0456 0.5mg (Experimental): oral
  Interventions: Drug: ASP0456
- Placebo group (Placebo Comparator): oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP0456 — oral
  Other Names: Linaclotide
  Arms: ASP0456 0.0625mg; ASP0456 0.125mg; ASP0456 0.25mg; ASP0456 0.5mg
Drug: Placebo — oral
  Arms: Placebo group

SUMMARY:
The objective of this study is to investigate dose-responses of efficacy and safety of ASP0456 in patients with chronic constipation (diagnosed by Rome III criteria of functional constipation (FC), not including constipation due to organic diseases) compared to placebo and to find the appropriate dose for P3 study.

DETAILED DESCRIPTION:
To determine optimum dose of ASP0456 for the patients with chronic constipation (not including constipation due to organic diseases) in Japan based on its efficacy and safety, multicentered, placebo-controlled, double-blind, parallel group comparative study will be conducted.

After two-week observation period, the patient who meets the primary registration criteria will be randomized to the one from five groups and will start treatment period. The patients will take once daily orally before the breakfast for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had SBM* (Spontaneous bowel movement) less than 3 times per week, more than six months prior to the provisional registration

  * *Defecation without procedure of laxative, suppository, enema, or stool extraction on the day or preceding day of the defecation
* Patient who was affected with one or more following symptoms before more than six months of provisional registration:

  * Straining during at least 25% of defecations
  * Lumpy or hard stools in at least 25% of defecations
  * Sensation of incomplete evacuation for at least 25% of defecations
* Loose stools are rarely present without the use of laxatives more than six months prior to the provisional registration.
* Patients who had pancolonoscopy or contrast enema (or sigmoidoscopy) after the onset of chronic constipation symptom and had no organic changes

Exclusion Criteria:

* Patient who has met IBS-C diagnostic criteria from Rome III more than six months prior to provisional registration. Meaning that patient who had recurrent abdominal pain or discomfort at least 3 days/month in last 3 months associated with two or more of the following, and patient who was affected with following IBS symptoms more than six months prior to the provisional registration:

  * Improvement with defecation
  * Onset associated with a change in frequency of stool
  * Onset associated with a change in form (appearance) of stool
* Patient with history of surgical resection of stomach, gallbladder, small intestine, or large intestine (excluding resection of appendicitis and benign polyp)
* Patient with history or current evidence of inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Patient with history or current evidence of ischemic colitis
* Patient currently affected by infectious enteritis
* Patient currently affected by hyperthyroidism or hypothyroidism
* Patient with apparent mechanical obstruction (i.e. patient with ileus caused by hernia)
* Patient with mega colon or mega rectum
* Patient currently affected by constipation due to anorectal dysfunction
* Patient currently affected by drug induced constipation.
* Patient with constipation due to other organic disease
* Patient currently affected by active peptic ulcer
* In the case of a female, the one currently affected by endometriosis or uterine adenomyosis
* Patient with high depression or anxiety considered to influence drug evaluation
* Patient with history of abuse of drug or alcohol within a year before consent acquisition, or with current abuse
* Patient who used or underwent or will use or undergo drug/therapy/test prohibited to combine 3 days before the start of bowel habit observation period (Day -17) or thereafter (however, patient who used or underwent restricted drug/therapy according to Protocol may be enrolled provisionally)
* Patient with history or current evidence of malignant tumor
* Patient currently affected by serious cardiovascular disease, respiratory disease, kidney disease, hepatic disease, gastrointestinal disease (excluding CC), hemorrhagic disease, or neural/mental disease
* Patient with history of drug allergy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Change in weekly average of SBM frequency | From baseline to week 1
  SBM: Spontaneous Bowel Movement. SBM means the defecation without procedure of laxative, suppository, enema, or stool extraction on the day or preceding day of the defecation. SBM frequency is calculated as follows: (the week total number of SBM )/ (the total number of days on which the frequency of SBM is evaluable) x7

SECONDARY OUTCOMES:
Weekly responder rate for SBM | up to 2 weeks
  The weekly average value of SBM frequency is more than 3 and over 1 more than the weekly mean value of SBM frequency in the bowel habit observation period
Weekly responder rate for CSBM | up to 2 weeks
  The weekly average value of CSBM frequency is more than 3 and over 1 more than the weekly mean value of CSBM frequency in the bowel habit observation period
Percentage of subjects with SBM within 24 hours after the start of initial treatment | up to 24 hours
Change in weekly average of CSBM frequency | From baseline to week 1
Proportion of subjects with CSBM within 24 hours after the start of initial treatment | up to 24 hours
Weekly responder rate of the global assessment of relief of chronic constipation. | up to 2 weeks
  The weekly responder of the evaluation items shall be the subject satisfying the following at the time of evaluation in each week: Score of Global assessment of relief of chronic constipation symptoms (7 scores: 1-7) is 1 or 2
Weekly responder rate of the abdominal bowel habits improvement in chronic constipation. | up to 2 weeks
  Score of abdominal bowel habits improvement effect (7 scores: 1-7) is 1 or 2
Weekly responder rate of abdominal symptom relief of chronic constipation. | up to 2 weeks
  Score of abdominal symptom improvement effect (7 scores: 1-7) is 1 or 2
Score of the global assessment of relief of chronic constipation | up to 2 weeks
  Scores will be measured using a seven-point ordinal score
Changes in IBS-QOL-J scores (entire scores or scores on the sub-scales) | Week 0, and 2
  IBS-QOL-J: Irritable bowel syndrome quality of life Japanese version
Changes in weekly average of SBM frequency | From baseline to every week until 2 weeks
  SBM: Spontaneous Bowel Movement
Changes in weekly average of CSBM frequency | From baseline to every week until 2 weeks
  CSBM: Complete Spontaneous Bowel Movement
Changes in weekly average of stool form | From baseline to every week until 2 weeks
  Stool form will be measured using seven-point Bristol Stool Form Scale
Changes in weekly average of abdominal bloating severity scores | From baseline to every week until 2 weeks
  Abdominal bloating severity will be measured using a five-point ordinal score
Changes in weekly average of abdominal pain/discomfort severity scores | From baseline to every week until 2 weeks
  Abdominal pain/discomfort severity will be measured using a five-point ordinal score
Changes in weekly average of straining severity scores | From baseline to every week until 2 weeks
  Straining severity will be measured using a five-point ordinal score
Score of the abdominal bowel habits improvement in chronic constipation | up to 2 weeks
  Scores will be measured using a seven-point ordinal score
Score of the abdominal symptom relief of chronic constipation | up to 2 weeks
  Scores will be measured using a seven-point ordinal score
Safety assessed by development of incidence of adverse events, vital signs, clinical laboratory tests and body weight | up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (50):
- Japan (50):
  - Site: 35, Aichi
  - Site: 36, Aichi
  - Site: 27, Chiba
  - Site: 28, Chiba
  - Site: 29, Chiba
  - Site: 30, Chiba
  - Site: 48, Fukuoka
  - Site: 49, Fukuoka
  - Site: 50, Fukuoka
  - Site: 1, Hokkaido
  - Site: 2, Hokkaido
  - Site: 45, Hyōgo
  - Site: 46, Hyōgo
  - Site: 47, Hyōgo
  - Site: 22, Kanagawa
  - Site: 23, Kanagawa
  - Site: 24, Kanagawa
  - Site: 25, Kanagawa
  - Site: 26, Kanagawa
  - Site: 44, Kyoto
  - Site: 37, Osaka
  - Site: 38, Osaka
  - Site: 39, Osaka
  - Site: 40, Osaka
  - Site: 41, Osaka
  - Site: 42, Osaka
  - Site: 43, Osaka
  - Site: 31, Saitama
  - Site: 32, Saitama
  - Site: 33, Saitama
  - Site: 34, Saitama
  - Site: 10, Tokyo
  - Site: 11, Tokyo
  - Site: 12, Tokyo
  - Site: 13, Tokyo
  - Site: 14, Tokyo
  - Site: 15, Tokyo
  - Site: 16, Tokyo
  - Site: 17, Tokyo
  - Site: 18, Tokyo
  - Site: 19, Tokyo
  - Site: 20, Tokyo
  - Site: 21, Tokyo
  - Site: 3, Tokyo
  - Site: 4, Tokyo
  - Site: 5, Tokyo
  - Site: 6, Tokyo
  - Site: 7, Tokyo
  - Site: 8, Tokyo
  - Site: 9, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Fukudo S, Miwa H, Nakajima A, Kinoshita Y, Kosako M, Nakagawa A, Akiho H, Kuroishi K, Johnston JM, Currie M, Ohkusa T. Dose-finding study of linaclotide in Japanese patients with chronic constipation: A phase II randomized, double-blind, and placebo-controlled study. Neurogastroenterol Motil. 2018 Dec;30(12):e13442. doi: 10.1111/nmo.13442. Epub 2018 Aug 7. PMID 30084233
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=279